CLINICAL TRIAL: NCT01068314
Title: Effect of Forearm Exercise on Flow Mediated Vasodilation Prior to Arteriovenous Fistula Placement for Hemodialysis
Brief Title: Effect of Exercise on Endothelial Function and Vascular Compliance in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Bradley S. Dixon, Associate Professor of Medicine, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UI200308021
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Kidney Failure, Chronic
Keywords: Endothelium; Vasodilatation; Vein; Compliance; Arteriovenous shunt, surgical
MeSH Terms: conditions — Kidney Failure, Chronic; Aneurysm; Patient Compliance; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Repetitive handgrip exercise (Experimental): After baseline testing and randomization, subjects in this group are instructed to perform the intervention: daily repetitive handgrip exercise with upper arm compression band. Brachial artery endothelial function and venous compliance are tested at baseline and 6 weeks.
  Interventions: Other: Repetitive arm exercise
- No arm exercise (No Intervention): Time control. Subjects do usual activities without any exercise intervention. Brachial artery endothelial function and venous compliance are tested at baseline and 6 weeks.

INTERVENTIONS:
Other: Repetitive arm exercise — After baseline testing and randomization, subjects in this group are instructed to perform repetitive handgrip exercise with an upper arm compression band until arm fatigue occurs. After resting 1 minute this exercise is repeated 9 times daily for 6 weeks.
  Arms: Repetitive handgrip exercise

SUMMARY:
The study hypothesis is that 6 weeks of repetitive handgrip exercise will improve endothelial function and venous compliance in pre-dialysis patients with an estimated glomerular filtration rate of less than or equal to 20 ml/min. If proven correct then arm exercise might be useful to improve the success rate for a surgically created arteriovenous fistula in the forearm to become usable as a vascular access for hemodialysis.

DETAILED DESCRIPTION:
An arteriovenous fistula (AVF) is the optimal vascular access for chronic hemodialysis. However, AVFs frequently fail to mature. Better strategies are needed to promote AVF maturation. Successful AVF maturation involves arterial and venous dilation. Arterial dilation depends on endothelial release of nitric oxide which can be measured by brachial artery flow-mediated dilation (FMD) and has been reported to predict successful AVF maturation. Venous dilation depends on venous compliance which can be measured by venous plethysmography and is also predictive of successful AVF maturation. Endothelial function is impaired in patients with chronic kidney disease (CKD). Aerobic exercise has been reported to improve endothelial function and venous compliance but it has not been studied in the pre-dialysis patient. To address this question we will determine whether 6 weeks of repetitive handgrip exercise with upper arm venous compression can improve brachial artery endothelial function or venous compliance in pre-dialysis patients with an estimated glomerular filtration rate of less than or equal to 20 ml/min.

ELIGIBILITY:
Inclusion Criteria:

* Age exceeding the age of majority (18 years of age).
* Chronic renal failure with a calculated GFR (MDRD equation) less than or equal to 20 ml/min
* Eligible for creation of an arteriovenous fistula for the purpose of hemodialysis.
* The subject is expected to stay within driving distance of study site for at least 4 months.
* The subject's physician(s) will allow the patient to participate.
* Ability to give informed consent.

Exclusion Criteria:

* Unstable angina.
* Uncontrolled hypertension (resting blood pressure >170 systolic or >100 diastolic).
* Musculoskeletal or neurologic problem that prevents arm exercise.
* Currently functioning arteriovenous access in the same arm as the planned new fistula.
* Subjects who are eligible to participate in the ongoing DAC fistula trial.
* Planned new access surgery in less than 6 weeks
* Anticipated non-compliance with medical care based on physician judgment.
* Patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilatation | 6 weeks

SECONDARY OUTCOMES:
Forearm venous compliance by plethysmography | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bradley S Dixon, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa General Clinical Research Center, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Nantakool S, Reanpang T, Prasannarong M, Pongtam S, Rerkasem K. Upper limb exercise for arteriovenous fistula maturation in people requiring permanent haemodialysis access. Cochrane Database Syst Rev. 2022 Oct 3;10(10):CD013327. doi: 10.1002/14651858.CD013327.pub2. PMID 36184076